CLINICAL TRIAL: NCT04468737
Title: Effect of Inadequate Bowel Preparation on Urgent Colonoscopy in Patients With Post-polypectomy Bleeding (PPB): A Descriptive Study
Brief Title: Effect of Inadequate Bowel Preparation on Urgent Colonoscopy in Patients With PPB.
Acronym: PPB
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PPB-1.0
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Post-polypectomy Bleeding; Bowel Preparation; Urgent Colonoscopy
MeSH Terms: interventions — Cathartics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Bowel preparation — Observe patients who undergo bowel preparation by enema or irrigation

SUMMARY:
The purpose of this study was to explore the effect of abbreviated bowel preparation on repeated colonoscopy in patients with PPB.

ELIGIBILITY:
Inclusion Criteria:

patients with bleeding after polypectomy patients treated with colonoscopy within 24 hours after bleeding patients who did not receive adequate bowel preparation (oral laxatives).

Exclusion Criteria:

patients whose main outcome indicators were not clearly described patients whose baseline characteristics were missing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing urgent colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic rate | 1 Day of colonoscopy
  the rate of identified the origin of the bleeding

SECONDARY OUTCOMES:
Ileocaecal intubation rate | 1 Day of colonoscopy
  the rate of colonoscopy entering the cecum

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China